CLINICAL TRIAL: NCT01049061
Title: A Phase 1 Study of MORAb-003 in Patients With Solid Tumor
Brief Title: A Study of MORAb-003 in Patients With Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MORAB-003-J081-102
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2014-02

CONDITIONS: Neoplasms; Solid Tumor
Keywords: Cancer; FRα
MeSH Terms: conditions — Neoplasms | interventions — farletuzumab

ARMS (1):
- MORAb-003 (Experimental)
  Interventions: Drug: MORAb-003

INTERVENTIONS:
Drug: MORAb-003 — MORAb-003 is intravenously administered to patients with solid tumor once a week for 4 weeks as 1 cycle in order to investigate dose-limiting toxicity and estimate maximum tolerated dose

SUMMARY:
MORAb-003 is intravenously administered to Japanese patients with folate receptor-alpha expressing solid tumor once a week for 4 weeks as 1 cycle in order to investigate dose-limiting toxicity and estimate maximum tolerated dose.

ELIGIBILITY:
Inclusion criteria;

1. Japanese male and female aged >or=20 to <80 years at obtaining informed consent
2. Patient with histologically or cytologically diagnosed solid tumor
3. Patient who is FRα-positive confirmed by immunohistochemistry (IHC) (except for ovarian cancer that FRα-positive is frequently reported)
4. Patients with a folate-receptor alpha expressing solid tumor who are not responsive or resistant to standard therapy and have no other appropriate treatment
5. Performance Status (PS) is 0 to 1 by Eastern Cooperative Oncology Group（ECOG）criteria

Exclusion criteria

1. Brain metastasis presenting clinical symptoms or requiring medical treatment
2. Serious and systemic infection requiring medical treatment
3. History of hypersensitivity to protein formulations including monoclonal antibody
4. With other active malignancy (except for carcinoma in situ)
5. With a large volume of pleural effusion or ascites requiring drainage

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To investigate dose-limiting toxicity and estimate maximum tolerated dose. | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chifumi Kitamura, Study Director — JAC PCU Eisai Co., Ltd.
Locations (2):
- Japan (2):
  - Hidaka-shi, Saitama
  - Chuo-ku, Tokyo

REFERENCES:
- [Derived] Sasaki Y, Miwa K, Yamashita K, Sunakawa Y, Shimada K, Ishida H, Hasegawa K, Fujiwara K, Kodaira M, Fujiwara Y, Namiki M, Matsuda M, Takeuchi Y, Katsumata N. A phase I study of farletuzumab, a humanized anti-folate receptor alpha monoclonal antibody, in patients with solid tumors. Invest New Drugs. 2015 Apr;33(2):332-40. doi: 10.1007/s10637-014-0180-8. Epub 2014 Nov 9. PMID 25380636